CLINICAL TRIAL: NCT00646490
Title: Diagnostic and Prognostic Values of Pleural Fluid Procalcitonin in Parapneumonic Pleural Effusion
Brief Title: Pleural Fluid and Serum Procalcitonin in Patients With Parapneumonic Pleural Effusion
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG840401
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2008-03

CONDITIONS: Community Acquired Pneumonia
Keywords: serum, pleural effusion, procalcitonin, pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia; Pleural Effusion; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum,pleural fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: patients with parapneumonic pleural effusion due to community acquired pneumonia
- B: patients with pleural effusion of other etiologies

SUMMARY:
Key words : serum, pleural effusion, procalcitonin, pneumonia Pneumonia is the common cause of pleural effusion (ranged 2nd) and bacterial infection is the main etiology of pneumonia. Procalcitonin, the prohormone of calcitonin, is a 116 amino-acid protein produced by C-cell of the thyroid gland. During severe infection, procalcitonin is probably produced by extra-thyroid tissues and the concentration increased rapidly in bacterial infection but remains low in viral infections. However, the exact origin and pathophysiological role of procalcitonin during sepsis is not clear and it is not a marker of infection as such, since localized infections or infections with no systemic manifestation cause a little if any increase in procalcitonin levels. This study will focus on assessing the value of procalcitonin in pleural effusion for diagnosis, severity and prognosis among community-acquired pneumonia with pleural effusion, such as in serum. 100 patients with clinical pneumonia infection score over six points diagnosed of community-acquired pneumonia and proved to have pleural effusion by chest sonography on admission will be studied prospectively. Serum and effusion procalcitonin levels will be measured initially and 3 days later after medical therapy. Bacterial pneumonia will be identified if bacteria was cultured from any one of the three kinds of specimen, including blood, pleural effusion or bronchoalveolar lavage. Then we will divide one hundred of patients into bacterial or non-bacterial groups. Finally, we will analyze demographic and procalcitonin data of serum and pleural effusion between these two groups and compare the difference between the severe or mild and response or non-response bacterial community-acquired pneumonia statistically.

The aim of the study will be to verify whether procalcitonin levels measured in the serum and pleural effusion could serve as a predictor for bacterial community-acquired pneumonia with pleural effusion and the different levels will also be indicative of severity and prognosis. We hope that the predictor from pleural effusion will be more sensitive or specific than that from serum and could be detectable in localized bacterial infection.

DETAILED DESCRIPTION:
In this study, the first goal will be to determine the sensitivity, specificity, and predictive value of serum and pleural effusion PCT level in CAP with pleural effusion. The second goal will be to decide an appropriate value in serum or pleural effusion to assess as an index of severity and prognosis in bacterial CAP with pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* A consecutive series of patients (17 years or older) who present to our hospital with suspected CAP with pleural effusion in the planning duration will be studied. All study cases had not received systemic or topical antimicrobial therapy during the 3 days before the study and they had never smoked at least one cigarette per day for 1 year. A case will be enrolled subsequently by the diagnosis of CAP with pleural effusion from clinical pneumonia infection score (CPIS) and chest sonography.

Exclusion Criteria:

* Patients with known thyroid disease or small cell lung cancer will be excluded.

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the out-patient-department in division of pulmonary and critical care medicine and the department of emergency medicine at Chang Gung Memorial Hospital, Kaohsiung.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2005-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
treatment response | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Chih Lin, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung, Kaohsiung City, Kaohsiung, Taiwan